CLINICAL TRIAL: NCT06619262
Title: The Effects of Concomitant Application of TENS and NMES on Chronic Stroke Patients: A Prospective Randomized Controlled Study
Brief Title: Concomitant Application of TENS and NMES on Chronic Stroke
Acronym: TENS NMES
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: After the G power analysis, it was determined that a total of 60 patients needed initial, 1st month and 4th month follow-ups. The study was terminated when the follow-ups of 60 patients were completed prospectively.
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Principal Investigator, Betül Başar, Assistant Professor, Gaziosmanpasa Research and Education Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Health Sciences
Record Dates: First submitted 2024-09-21; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Stroke; Hemiparesis
Keywords: Stroke; Exercise program; TENS; NMES
MeSH Terms: conditions — Stroke; Paresis | interventions — Transcutaneous Electric Nerve Stimulation; Resistance Training

STUDY DESIGN:
Intervention Model Description: This is a prospective randomized assessor-blind comparison study.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- TENS+NMES Group (Experimental): The group in which TENS and NMES are applied concomitantly in the treatment
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Device: Neuromuscular and Muscular Electrical Stimulation; Other: Exercise program
- TENS Group (Active Comparator): The group in which TENS is applied concomitantly in the treatment
  Interventions: Device: Transcutaneous Electrical Nerve Stimulation; Other: Exercise program
- NMES Group (Active Comparator): The group in which NMES is applied concomitantly in the treatment
  Interventions: Device: Neuromuscular and Muscular Electrical Stimulation; Other: Exercise program
- Control (Sham Comparator): No additional electrical stimulation is applied for treatment in this group.
  Interventions: Other: Exercise program

INTERVENTIONS:
Device: Transcutaneous Electrical Nerve Stimulation — TENS stands for transcutaneous electrical nerve stimulation. Transcutaneous means across the skin. TENS machines pass a small electrical current across your skin to stimulate the nerves.
  Arms: TENS Group; TENS+NMES Group
Device: Neuromuscular and Muscular Electrical Stimulation — Neuromuscular and Muscular Electrical Stimulation (NMES) is a modality that sends electrical impulses to nerves which causes the muscles to contract mimicking the action potential coming from the central nervous system.
  Arms: NMES Group; TENS+NMES Group
Other: Exercise program — Specific exercise program for patients with lower extremity hemiparesis after stroke

SUMMARY:
Stroke is a cerebrovascular disorder that can lead to permanent disability and a decline in quality of life. Chronic stroke patients often experience decreased balance control, which negatively affects activities of daily living and their ability to walk independently. Studies conducted with electrical stimulation have shown that it is safe to use on humans. Today, it is frequently preferred in treatment.

Electrical stimulation are effective for treatment of stroke. Electrical stimulation has been used as transcutaneous nerve stimulation (TENS) and neuromuscular electrical stimulation (NMES). Both of them are effective but not sufficient. The concomitant application of TENS and NMES may achieve better results than individually application.

DETAILED DESCRIPTION:
Stroke is a cerebrovascular disorder that can lead to permanent disability and a decline in quality of life. Chronic stroke patients often experience decreased balance control, which negatively affects activities of daily living and their ability to walk independently. The most recognized impairments are deficits in motor control and limited mobility. Chronic stroke patients may develop spasticity, which is the main cause of decreased balance and gait. The rate of post-stroke spasticity is 4 - 27% in the 6th week, increasing to 42.6% by the 6th month. Electrical stimulation has been used in numerous studies to decrease spasticity.

Electrical stimulation has been widely used in stroke rehabilitation, including transcutaneous nerve stimulation (TENS) and neuromuscular electrical stimulation (NMES). NMES is an effective and conventional therapeutic method for improving motor function in patients with lower extremity paralysis after stroke. During NMES, current pulses are applied to the muscles or motor nerves through surface electrodes to induce muscle contractions to mimic exercise therapy. NMES can help improve muscle strength, joint range of motion, and promote motor relearning. TENS, another electrical stimulation, is used to relieve pain, improve muscle strength and motor function, and reduce spasticity through transdermal output pulses. The motor recovery mechanism of TENS involves the presynaptic inhibition of the hyperactive stretch reflexes in spastic muscles and decreased co-contraction of the spastic antagonist muscles.

Numerous studies have investigated the benefits of TENS or NMES applied to the lower extremities. These studies have revealed that both forms of electric stimulation are effective in the recovery of chronic stroke patients.

However, there is no comparative study on the effect of TENS and NMES applied individually versus their concomitant application. The combined application of TENS and NMES may yield better results. The aim of this study is to compare the effects of TENS and NMES, applied both individually and concomitantly, on posture, lower extremity motor recovery, functional independence, motor function recovery, and spasticity. Hypothesis is that the concomitant application of TENS and NMES will achieve better results than individually application.

ELIGIBILITY:
Inclusion Criteria:

First episode of unilateral stroke with hemiparesis Stroke confirmed by CT and/or MRI Ablity to independently stand up from a chair

Exclusion Criteria:

Cerebellar or brainstem stroke Severe cognitive and communication impairment Previous surgical treatment history on the affected extremity Complication with severe heart, lung, liver, kidney, or infectious disease Presence of a cardiac pacemaker Orthopedic disease affecting sit-to-stand movement Inability to understand and follow verbal commands Peripheral or central nervous system dysfunction

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale | up to 4 months
  Disability caused by stroke was evaluated using the National Institutes of Health Stroke Scale (NIHSS). The following domains were assessed with the NIHSS: level of consciousness, eye movements, integrity of visual fields, facial movements, arm and leg muscle strength, sensation, coordination, language, speech and neglect. Evaluation was based on a total score ranging from 0 to 42, with higher the scores indicating more severe stroke.
Brunnstrom's Hemiplegia Recovery Staging | up to 4 months
  The lower extremity motor recovery was assessed using Brunnstrom's Hemiplegia Recovery Staging. There are six grades in Brunnstrom's Hemiplegia Recovery Staging for the lower extremity. A higher stage indicates better motor function. The Brunnstrom stages were preferred because they reflect the underlying motor control based on clinical assessment of movement quality.
Postural Assessment Scale for Stroke Patients | up to 4 months
  Postural Assessment Scale for Stroke Patients (PASS) was developed specifically for evaluating balance in stroke patients. PASS contains two subheadings for evaluating balance: maintaining posture (static PASS) and changing posture (dynamic PASS). It consists of 12 items to evaluate balance: 5 items (sitting without support; standing with support; standing without support; standing on the non-paretic leg; standing on the paretic leg) for static PASS, and 7 items (supine to affected side lateral; supine to non-affected side lateral; supine to sitting up on the edge of the mat; sitting on the edge of the mat to supine; sitting to standing; standing to sitting down; standing, picking up a pencil from the floor) for dynamic PASS. Evaluation was based on a total score ranging from 0 to 36, with higher the scores indicating more favorable balance in stroke patients.
Functional Independence Measures | up to 4 months
  Functional Independence Measures (FIM) is widely used to assess the independence of stroke patients. It contains 18 items under the following categories: self-care, sphincter control, transfers, locomotion, communication and social cognition. Each item was scored from 1 to 7, with 7 indicating complete independence and 1 indicating complete dependence. Scores below 6 indicate that the patient requires assistance or supervision from another person.
Modified Ashworth Scale | up to 4 months
  The Modified Ashworth Scale (MAS) was used to assess the spasticity of the ankle plantar flexors. The physiotherapist passively moved the ankle from maximal plantarflexion to maximal dorsiflexion. The MAS assigns a grade of spasticity on a scale of 0-4 based on the level of resistance in response to passive movement. A score of 0 represents no increase in muscle tone, while a score of 4 represents rigidity of the affected part in flexion or extension.

SECONDARY OUTCOMES:
Electrical stimulation side effects | up to 4 months
  Skin lesions, muscle cramps or ruptures, and neurovascular side effects that may occur with the combined application of TENS and NMES will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Basar B, Alp OF. The effects of concomitant application of TENS and NMES on chronic stroke patients: a prospective randomized controlled study. BMC Sports Sci Med Rehabil. 2025 Apr 24;17(1):91. doi: 10.1186/s13102-025-01155-w. PMID 40275398